CLINICAL TRIAL: NCT02624674
Title: Multi-spectral Imaging to Assess Wounds in Peripheral Vascular Disease Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-249c
Record Dates: First submitted 2015-08-13; First posted 2015-12-08 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Peripheral Vascular Disease Patient
MeSH Terms: interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Multi-spectral Imaging Group (Experimental): All subjects in this group will undergo baseline Near Infrared Spectroscopy (NIRS) measurement points with the Multi-spectral imaging device, baseline vascular studies (including ankle-brachial index (ABI), vascular doppler (arterial and venous), and toe pressures. At the one month mark (from baseline), NIR measurement point and vascular studies will again be performed. All measurements are incorporated into the routine wound care and will not require extra trips in hospital for wound care.
  Interventions: Device: Multi-spectral Imaging Device (MSID)

INTERVENTIONS:
Device: Multi-spectral Imaging Device (MSID)
  Other Names: Near infrared spectroscopy (NIRS)

SUMMARY:
Peripheral vascular disease (PVD) is a common disease of impaired blood flow resulting in the compromised tissue perfusion of lower limbs. PAD patients can experience pain, diminished exercise capacity, and tissue loss, with some ultimately requiring amputation. The economic burden of PVD is significant. In the United States alone, PVD accounts for over $20 billion in annual healthcare related costs.

The demand for the development of an effective method to characterize the viability of PVD wounds has resulted in the emergence of several innovative techniques. Commonly used diagnostic methods are ankle-brachial index (ABI), pulse volume recordings, duplex ultrasonography, venous plethysmography, Transcutaneous oxygen tension (TcPO2), toe pressures, angiography by X-ray, computed tomography, and magnetic resonance imaging. Currently, angiography remains the diagnostic gold standard. However, many of these techniques lack the ability to triage and adequately determine the viability of the wound. In addition, there remains a need for effective triage technologies to help clinicians decide whether surgical management is needed. Early determination of surgical versus conservative management may help to improve patient functional outcomes, reduce mortality rates, and prevent limb amputation.

Near-infrared point spectroscopy (NIRS) is a non-invasively technology with recent applications in PVD wound assessment. To date, studies have demonstrated the validity of NIRS technology in patients with peripheral arterial disease. NIRS measures flow, concentration, and oxygenation of hemoglobin in arterioles, capillaries, and venules several centimeters deep in tissue. The MSID is an evolution of existing NIRS imaging devices and has become a portable and functional commercial device produced by KENT imaging (Calgary, Canada). Using this new and clinically applicable NIRS technology designed for assessing wound perfusion and oxygenation, this study seeks to adequately identify viable from non-viable wounds and to rapidly determine indication for vascular interventions. This technology is well-suited for use in a wound patient population as the measurements times are short and can quickly be used at the patient bed side. As such, this project intends to apply NIR technology to quickly assess PVD in the investigators' patient population.

DETAILED DESCRIPTION:
Peripheral vascular disease (PVD) is a common disease of the elderly, resulting in the compromise of blood flow to the lower limbs. As a consequence of impaired tissue perfusion, PAD patients can experience pain, diminished exercise capacity, and tissue loss, with some ultimately requiring amputation. Globally, lower extremity peripheral artery disease is the third leading cause of atherosclerotic cardiovascular morbidity, affecting over 200 million individuals worldwide. Peripheral vascular disease is becoming more prevalent with the increase of incidence with age and a globally aging population. In 2010, it was estimated that the number of people living with peripheral artery disease increased by 23.5% in the last decade. The economic burden of PVD is significant. In the United States alone, PVD accounts for over $20 billion in annual healthcare related costs. Specifically, non-healing wounds represent a significant portion of this expenditure at more than $3 billion per year.

The demand for the development of an effective method to characterize the viability of PVD wounds has resulted in the emergence of several innovative techniques. Commonly used diagnostic methods are ankle-brachial index (ABI), pulse volume recordings, duplex ultrasonography, venous plethysmography, angiography by X-ray, computed tomography, and magnetic resonance imaging. However, many of these techniques lack the ability to triage and adequately determine the viability of the wound. Ankle brachial index (ABI) is one of the most common screening techniques used to establish the presence of PVD, but it lacks sensitivity in creating sensitive and specific categorization of wounds as viable or non-viable. ABI gives an indication of a hemodynamically significant obstruction, but does not measure blood flow directly. Doppler ultrasound is another common method that can measure arterial blood flow, however some groups suggest that the femoral artery blood flow may not be an accurate hemodynamic indication of muscle ischemia. Magnetic resonance spectroscopy is also a new technique that has been validated in its application to assess PVD. Novel magnetic imaging sequences such as PIVOT (Perfusion, Intravascular Venous Oxygen Saturation) combine Blood Oxygen Level Dependent (BOLD) MRI and Arterial Spin Labeling (ASL) to comprehensively assess the tissue. Despite the strengths that many MRI techniques promise, clinical use limitations remain due to the high costs and availability of resources.

Peripheral vascular disease-induced lower extremity wounds have inadequate perfusion. Currently, there are three major approaches to improve vascular perfusion to the area: medical management, open surgery, and endovascular surgery. Medical management consists of lifestyle modification and management of associated risk factors such as smoking, diabetes mellitus, hyperlipidemia, hypertension, and hypercoagulability. While advances have been made in the medical management of lower extremity ischemia-induced wounds, large arterial revascularization remains the current standard of care. Open bypass surgery is often employed to bypass stenotic arteries and improve perfusion to lower extremity wounds. Over the last two decades, endovascular intervention has emerged as an additional therapy as it is minimally invasive and may have lower associated morbidity and mortality. In addition to improved perfusion of lower extremity wounds by medical management of surgical intervention, local wound care is required to expedite the healing process and prevent infection.

However, there remains a need for effective triage technologies to help clinicians decide whether surgical management is needed. This would allow for early determination of surgical versus conservative management and inpatient versus outpatient management. If surgery is required, patient functional outcomes are improved if it takes place earlier. As well, inpatient management of surgical patients is extremely costly. Outpatient management of patients with peripheral vascular wounds that do not require surgery would significantly reduce the costs associated with surgical intervention.

Near-infrared point spectroscopy (NIRS) non-invasively measures flow, concentration, and oxygenation of hemoglobin in arterioles, capillaries, and venules several centimeters deep in tissue. NIRS is safe and comfortable for patients and is well-suited to measure markers of viability in peripheral vascular disease wounds, including tissue perfusion, oxygenation and hemoglobin. To date, studies have demonstrated the validity of NIRS technology in patients with peripheral arterial disease. The Multi spectrum infrared device (MSID) represents an important evolution of existing NIRS imaging devices, which were designed for the clinical environment. The MSID has become a commercial device produced by KENT imaging (Calgary, Canada) after several animal and clinical trials have validated its use. The MSID is a new generation of NIR imaging devices with enhanced portability and functionality. The MSID is able to monitor many variables, such as cytochrome oxidase as a marker of tissue oxygen utilization, oxygen saturation, perfusion and methemoglobin as a marker of free radical injury. The advantage of the MSID is its capacity to account for skin colour. Melanin absorbs light and attenuates the amount of NIR light received by the camera. The Kent imaging device has unique mathematical algorithms to account for melanin content of the skin. In many previous studies done with NIRS technology in PVD wounds, melanin content was not considered to be a factor as patients demographic was predominantly Caucasian. However, in many multicultural cities where there is a wide variability in patient melanin content, melanin corrections in NIRS imaging are very important.

Using this new and clinically applicable NIRS technology designed for PVD, this study seeks to identify viable from non-viable wounds and to determine the severity of wound in assessing for vascular intervention indication. This technology is well-suited for use in a wound patient population as the measurements times are short and movement of subjects is not an issue. As such, this project intends to apply novel technology that has the capacity to quickly assess wounds as a complication of PVD.

ELIGIBILITY:
Inclusion Criteria

1. Lower extremity wound from peripheral vascular disease, which has had optimum multi-disciplinary team management for >4 weeks
2. Wound size of <10 cm
3. In-patients or out-patients in the care of St.Michael's Hospital (SMH) wound care team
4. Patients aged >18 years
5. Patients who understand the study, agree to adhere to the treatment and are able to give consent
6. Patients who can be followed by the same investigating team for the whole period of their participation in the study

3.3 Exclusion Criteria

1. Presence of invasive infection requiring intravenous antibiotics or debridement.
2. Significant reduced immunity or high dose corticosteroids (>10mg Prednisolone) or other second line immune-suppressant
3. Need for total contact cast
4. Patients with known or suspected malignancy in the wound or surrounding tissue.
5. Patients who are participating in another clinical study for peripheral vascular diseae wound management
6. Patients with a known history of poor compliance with medical treatment
7. Foot wounds
8. Diabetic patients who cannot have reliable ABI measurements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in ABI (scale measurement) | 1 month
  The Ankle-brachial index (ABI) result is used to predict the severity of peripheral vascular disease (PVD). The ankle-brachial index test compares blood pressure measured at the ankle with the blood pressure measured at the arm. ABI is measured on a scale from <0.5 to >1.5
Change from baseline in Vascular Doppler (imaging analysis) | 1 month
  Doppler ultrasound is a special ultrasound technique that uses sound waves to non-invasively evaluate the blood flow through arteries and veins in the body. Blood flow measurements from vascular doppler are measured in mL/min.
Change from baseline in Toe pressures (physiological parameter measurement) | 1 month
  Toe pressures are non-invasive blood pressure measurements taken at the toe and measured in mmHg.
Change from baseline in Angiography (imaging analysis) | 1 month
  Angiography or arteriography is a x-ray medical imaging technique used to visualize the inside (lumen) of blood vessels and organs in the body. Analysis is given by imaging experts (i.e., radiologists, cardiologists, or technologists) in a descriptive report.
Change from baseline in Oxygen saturation from the MSID device (scale measurement) | 1 month
  Using visible and near infrared light, oxygen saturation can non-invasively be determined from using the MSID device. Oxygen saturation is measured in percentage from 0-100%.
Change from baseline in Total hemoglobin from the MSID device (physiological parameter measurement) | 1 month
  Using visible and near infrared light, total hemoglobin can non-invasively be determined from using the MSID device. Total hemoglobin is measured by g/L.
Change from baseline in Wound Healing (physiological parameter measurement) | 1 month
  Wound healing is determined by the amount of change in the wound surface area (measured in mm^2)

REFERENCES:
- [Background] Kramer CM. Skeletal muscle perfusion in peripheral arterial disease a novel end point for cardiovascular imaging. JACC Cardiovasc Imaging. 2008 May;1(3):351-3. doi: 10.1016/j.jcmg.2008.03.004. PMID 19356448
- [Background] Fowkes FG, Rudan D, Rudan I, Aboyans V, Denenberg JO, McDermott MM, Norman PE, Sampson UK, Williams LJ, Mensah GA, Criqui MH. Comparison of global estimates of prevalence and risk factors for peripheral artery disease in 2000 and 2010: a systematic review and analysis. Lancet. 2013 Oct 19;382(9901):1329-40. doi: 10.1016/S0140-6736(13)61249-0. Epub 2013 Aug 1. PMID 23915883
- [Background] McDermott MM. Peripheral arterial disease: epidemiology and drug therapy. Am J Geriatr Cardiol. 2002 Jul-Aug;11(4):258-66. doi: 10.1111/j.1076-7460.2002.00031.x. PMID 12091774
- [Background] Menke NB, Ward KR, Witten TM, Bonchev DG, Diegelmann RF. Impaired wound healing. Clin Dermatol. 2007 Jan-Feb;25(1):19-25. doi: 10.1016/j.clindermatol.2006.12.005. PMID 17276197
- [Background] Bernink, P. J. L. M., Lubbers, J., Barendsen, G. J., and Van den try in the assessment of peripheral arterial disease. Adv. Exp.
- [Background] Lewis P, Psaila JV, Morgan RH, Davies WT, Woodcock JP. Common femoral artery volume flow in peripheral vascular disease. Br J Surg. 1990 Feb;77(2):183-7. doi: 10.1002/bjs.1800770220. PMID 2317678
- [Background] Zatina MA, Berkowitz HD, Gross GM, Maris JM, Chance B. 31P nuclear magnetic resonance spectroscopy: noninvasive biochemical analysis of the ischemic extremity. J Vasc Surg. 1986 Mar;3(3):411-20. doi: 10.1067/mva.1986.avs0030411. PMID 2936903
- [Background] Kramer CM. Novel magnetic resonance imaging end points for physiologic studies in peripheral arterial disease: elegance versus practicality. Circ Cardiovasc Imaging. 2015 Apr;8(4):10.1161/CIRCIMAGING.115.003360 e003360. doi: 10.1161/CIRCIMAGING.115.003360. No abstract available. PMID 25873725
- [Background] Bunte MC, Shishehbor MH. Treatment of infrapopliteal critical limb ischemia in 2013: the wound perfusion approach. Curr Cardiol Rep. 2013 Jun;15(6):363. doi: 10.1007/s11886-013-0363-5. PMID 23605465
- [Background] Romiti M, Albers M, Brochado-Neto FC, Durazzo AE, Pereira CA, De Luccia N. Meta-analysis of infrapopliteal angioplasty for chronic critical limb ischemia. J Vasc Surg. 2008 May;47(5):975-981. doi: 10.1016/j.jvs.2008.01.005. Epub 2008 Apr 18. PMID 18372148
- [Background] Cross, K. M. 2010. Assessing tissue viability of acute thermal injuries using near infrared point spectroscopy.
- [Background] Cross KM, Leonardi L, Gomez M, Freisen JR, Levasseur MA, Schattka BJ, Sowa MG, Fish JS. Noninvasive measurement of edema in partial thickness burn wounds. J Burn Care Res. 2009 Sep-Oct;30(5):807-17. doi: 10.1097/BCR.0b013e3181b485e9. PMID 19692905
- [Background] Cross KM, Leonardi L, Payette JR, Gomez M, Levasseur MA, Schattka BJ, Sowa MG, Fish JS. Clinical utilization of near-infrared spectroscopy devices for burn depth assessment. Wound Repair Regen. 2007 May-Jun;15(3):332-40. doi: 10.1111/j.1524-475X.2007.00235.x. PMID 17537120
- [Background] Leonardi L, Sowa MG, Payette JR, Mantsch HH. Near-infrared spectroscopy and imaging: a new approach to assess burn injuries. Am Clin Lab. 2000 Sep-Oct;19(8):20-2. No abstract available. PMID 11146988
- [Background] Sowa MG, Leonardi L, Payette JR, Cross KM, Gomez M, Fish JS. Classification of burn injuries using near-infrared spectroscopy. J Biomed Opt. 2006 Sep-Oct;11(5):054002. doi: 10.1117/1.2362722. PMID 17092151
- [Background] Sowa MG, Leonardi L, Payette JR, Fish JS, Mantsch HH. Near infrared spectroscopic assessment of hemodynamic changes in the early post-burn period. Burns. 2001 May;27(3):241-9. doi: 10.1016/s0305-4179(00)00111-x. PMID 11311517
- [Background] Cheatle TR, Potter LA, Cope M, Delpy DT, Coleridge Smith PD, Scurr JH. Near-infrared spectroscopy in peripheral vascular disease. Br J Surg. 1991 Apr;78(4):405-8. doi: 10.1002/bjs.1800780408. PMID 2032098
- [Background] Komiyama T, Shigematsu H, Yasuhara H, Muto T. An objective assessment of intermittent claudication by near-infrared spectroscopy. Eur J Vasc Surg. 1994 May;8(3):294-6. doi: 10.1016/s0950-821x(05)80144-6. PMID 8013679
- [Background] Komiyama T, Shigematsu H, Yasuhara H, Muto T. Near-infrared spectroscopy grades the severity of intermittent claudication in diabetics more accurately than ankle pressure measurement. Br J Surg. 2000 Apr;87(4):459-66. doi: 10.1046/j.1365-2168.2000.01381.x. PMID 10759743
- [Background] Egun A, Farooq V, Torella F, Cowley R, Thorniley MS, McCollum CN. The severity of muscle ischemia during intermittent claudication. J Vasc Surg. 2002 Jul;36(1):89-93. doi: 10.1067/mva.2002.123678. PMID 12096263